CLINICAL TRIAL: NCT02756026
Title: Assessing the Quality of Breast Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BMQ; 429296-1 (Other: University of California, Davis)
Record Dates: First submitted 2016-04-13; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Micronutrient Deficiency
Keywords: Breast milk; mineral; vitamin
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micronutrient supplementation (Experimental): On day 3, all mothers are given a commercial multiple micronutrient supplement (Nutri-Fem) manufactured by Thorne, containing the Recommended Dietary Intake (RDA).
  On day 4, all mothers are given two commercial multiple micronutrient supplements (Nutri-Fem) manufactured by Thorne, containing twice the Recommended Dietary Intake (RDA).
  Interventions: Dietary Supplement: Multiple micronutrient supplement (Nutri-Fem)

INTERVENTIONS:
Dietary Supplement: Multiple micronutrient supplement (Nutri-Fem) — Multiple micronutrient supplement (Nutri-Fem) manufactured by Thorne, containing the Recommended Dietary Intake (RDA).

SUMMARY:
The purpose of the study is to establish a protocol for collecting representative samples of breastmilk (BM) that can be used to assess the effect of maternal micronutrient (MN) supplementation on milk MN concentrations. The investigators will determine which breastfeeding episode during the 24 hour period best represents the maternal status; and within the episode whether fore, mid or hind milk samples be collected in future studies.

DETAILED DESCRIPTION:
Mother-infant pairs were recruited in the peri urban area of Dhaka, Bangladesh to participate in a protocol development study at International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b). The participants will spend 5 days in a metabolic unit of icddr,b and the procedures are as follows:

* On day 1, mother-infant pairs will come to the facility, consume their evening meal and spend the night.
* On day 2, the mothers will be asked to breastfeed their infant from one breast for as long as the infant is interested. An electric breast pump will be placed simultaneously on the other breast for a Full Milk (FM) collection. For the duration of the study the same breast will be used for feeding the infant the other breast will be used for the FM collection. Three separate aliquots of fore milk (up to 1 minute), mid (50 mL), and hind (until the breast is empty) milk will be collected by a special funnel attached to the breast pump. A 5 mL aliquot of BM will be removed from each the 3 aliquots for creamatocrit measurement and later vitamin and mineral determinations. The remainder of the pumped breast milk will be pooled and given to the mother to feed to her infant. A fasting blood sample (7 mL) will be obtained by venipuncture to measure maternal MN status. A breakfast meal will be served to the mother after the first feeding and the blood draw. The mother will be asked to refrain from breastfeeding her infant for the next 2-3 hours then the collection procedure will be repeated until the mother goes to sleep at night, and at any time during the night that the mother wakes to feed her infant. The meals for breakfast, lunch and dinner will be low in micronutrients.
* On day 3, the mothers will be given one commercial multiple micronutrient supplement tablet containing the Recommended Dietary Intake (RDA). Milk collection procedures will be repeated the same as on day 2. The meals for breakfast, lunch and dinner will be low in micronutrients. Between breast milk collections the staff will collect maternal and infant anthropometry data, and administer Food Frequency (FF) and morbidity questionnaires.
* On day 4, the mothers will be given two commercial multiple micronutrient supplement tablets containing the Recommended Dietary Intake (RDA). Milk collection procedures will be repeated the same as on day 3. The meals for breakfast, lunch and dinner will be low in micronutrients.
* On day 5, the study will end with a final collection of BM in the morning and the study participants will be discharged from the facility.

ELIGIBILITY:
Inclusion Criteria:

* BMI >18.5 Healthy
* In the 2nd to 4th month of lactation and breastfeeding ≥12 times/d
* Breast-feeding only one infant
* Non-pregnant
* Willing to spend 4 days and nights at the metabolic unit
* Willing to perform the procedures of BM collection using the breast pump.

Exclusion Criteria:

* Severe anemia (Hb <90 g/L) by HemoCue
* Currently taking micronutrient supplements
* Current pregnancy
* Current illness
* Current Mastitis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in Breast Milk Content of Cobalamin (Vitamin B12) | Breast milk is collected at every infant feeding on days 2, 3 and 4 and is divided into fore, mid and hind milk
  Vitamin B12 (ng/L) is measured in breast milk by quantitative immunoassay

SECONDARY OUTCOMES:
Plasma Cobalamin (Vitamin B12) | Measured once in a fasting blood sample collected on day 2
  Vitamin B12 (pmol/L) is measured in plasma by automated immunoassay
Plasma Folate | Measured once in a fasting blood sample collected on day 2
  Folate (nmol/L) is measured in plasma by automated immunoassay
Change in Breast Milk Content of Thiamin | Breast milk is collected at every infant feeding on days 2, 3 and 4 and is divided into fore, mid and hind milk
  Thiamin in breast milk (ug/L) is measured as Thiamin, Thiamin-monophosphate, and Thiamin-pyrophosphate by high performance liquid chromatography (HPLC)
Change in Breast Milk Content of Riboflavin | Breast milk is collected at every infant feeding on days 2, 3 and 4 and is divided into fore, mid and hind milk
  Riboflavin in breast milk (ug/L) is measured as Riboflavin and Flavin adenine dinucleotide by ultra-performance liquid chromatography followed by tandem mass spectrometry (UPLC-MS/MS)
Change in Breast Milk Content of Niacin | Breast milk is collected at every infant feeding on days 2, 3 and 4 and is divided into fore, mid and hind milk
  Niacin in breast milk (ug/L) is measured as Nicotinamide by UPLC-MS/MS
Change in Breast Milk Content of Vitamin B6 | Breast milk is collected at every infant feeding on days 2, 3 and 4 and is divided into fore, mid and hind milk
  Vitamin B6 in breast milk (ug/L) is measured as Pyridoxal by UPLC-MS/MS
Change in Breast Milk Content of Vitamin A | Breast milk is collected at every infant feeding on days 2, 3 and 4 and is divided into fore, mid and hind milk
  Vitamin A in breast milk (nmol/L) is measured as retinol and beta-carotene by HPLC
Change in Breast Milk Content of Vitamin E | Breast milk is collected at every infant feeding on days 2, 3 and 4 and is divided into fore, mid and hind milk
  Vitamin E in breast milk (nmol/L) is measured as alpha-tocopherol and gamma-tocopherol by HPLC
Change in Breast Milk Content of fat | Breast milk is collected at every infant feeding on days 2, 3 and 4 and is divided into fore, mid and hind milk
  Fat in breast milk (g/L) is measured using a creamatocrit.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay H Allen, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hampel D, Shahab-Ferdows S, Islam MM, Peerson JM, Allen LH. Vitamin Concentrations in Human Milk Vary with Time within Feed, Circadian Rhythm, and Single-Dose Supplementation. J Nutr. 2017 Apr;147(4):603-611. doi: 10.3945/jn.116.242941. Epub 2017 Feb 15. PMID 28202638